CLINICAL TRIAL: NCT04029883
Title: Behavioral Economics to Improve Antihypertensive Therapy Adherence (BETA)
Brief Title: Behavioral Economics to Improve Antihypertensive Therapy Adherence
Acronym: BETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: RAND (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph Ebinger, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00057764; 1R21HL156132-01 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Medication Adherence
Keywords: hypertension; medication adherence; behavioral economics
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The Control group will receive care as usual, as well as a MEMS-cap and a leaflet explaining the importance of pill-taking routines and how to establish them. The study coordinator will spend approximately ten minutes with them to go over the leaflet and answer questions. Control group participants also spend time with the study coordinator at each clinic visit where contact information is updated, and any MEMS-cap problems are resolved. These procedures, which we successfully applied in previous studies, minimize the possibility that results are confounded by differences in attention or other non-specific effects between groups.
- Message Group (Active Comparator): The Message group will receive the same brief information session as the Control group but also receive daily text messages reinforcing the information provided for 3 months. A key insight from BE is that people typically are initially highly motivated to change their behavior, but their enthusiasm declines over time. To keep the importance of routinizing pill- taking salient (i.e. high on a person's mental priority list), we will send daily text messages using a freely available web platform. These messages will reinforce the information provided at recruitment, and remind participants of their personalized routinization strategy. Messages will be tailored and refreshed based on patient-specific factors including BP control, prior adherence, and current medication regimen.
  Interventions: Behavioral: Text Message
- Incentive Group (Experimental): The Incentive group will receive the same information and text messages, but in addition have a chance of winning small, intermittent rewards for taking their medication at the time coinciding with their anchoring strategy. In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits. When the participants return for their monthly visit, the study coordinator will download their MEMS-cap data and check whether this eligibility criteria was satisfied. MEMS software can be easily customized to display this information. If the patient qualifies, s/he is invited to draw one of three laminated cards with numbers 0, 25, and 50 out of a bag. The client receives the corresponding amount in USD in the form of a gift card immediately after the drawing.
  Interventions: Behavioral: Behavior Economic Incentive; Behavioral: Text Message

INTERVENTIONS:
Behavioral: Text Message — A key insight from BE is that people typically are initially highly motivated to change their behavior, but their enthusiasm declines over time.103 To keep the importance of routinizing pill-taking salient (i.e. high on a person's mental priority list), we will send daily text messages using a freely available web platform.
  Arms: Message Group
Behavioral: Behavior Economic Incentive — In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits.
  Arms: Incentive Group
Behavioral: Text Message — A key insight from BE is that people typically are initially highly motivated to change their behavior, but their enthusiasm declines over time.103 To keep the importance of routinizing pill-taking salient (i.e. high on a person's mental priority list), we will send daily text messages using a freely available web platform.
  Arms: Incentive Group

SUMMARY:
Hypertension represents a major cardiovascular risk factor that can be controlled through the use of medications, yet medication non-adherence represents a common problem that leaves patients at elevated risk for adverse cardiovascular outcomes. Interventions to improve medication adherence have thus far been either unsuccessful or unsustainable. The investigators propose an intervention that leverages insights from behavioral economics to improve medication adherence among hypertensive patients. Strong data indicates that linking the taking of medications to daily routines ('anchoring') increases adherence, however, existing interventions built on this information have failed to create successful, long term improvements in medication adherence. This study aims to leverage behavioral economic insights to improve medication adherence to antihypertensive medications.

DETAILED DESCRIPTION:
The investigators propose to complement linking medication taking to a daily routine with two added components to make it easier for participants to stick to their anchoring plan: increasing information salience through frequent text messages and providing intermittent rewards for pill-taking according to the anchoring plan.

This study will be implemented in a pilot randomized controlled trial (RCT) in a high-volume clinical practice to establish feasibility, acceptability, and preliminary efficacy. The specific aims include 1) a formative phase to develop the intervention and evaluate its feasibility and acceptability via focus groups with key stakeholders; 2) a RCT of 60 hypertensive patients in which a control group (n=20) is provided education on anchoring medication taking to a daily routine, and two intervention groups, one (n=20) who receives anchoring education and daily text message reminders and another (n=20) which receives anchoring education, text messages, and financial incentives for adherence in accordance with their anchoring plan; and 3) data collection in preparation for a future R01 application, including focus group discussions with key stakeholders (patients, providers [Physicians, Nurses, Advanced Care Practitioners, Pharmacists] and clinic staff) and exit focus groups with study participants regarding ways to improve the intervention.

The main hypothesis is: the intervention is effective by anchoring pill-taking to an existing routine, tested by comparing the pooled (Message group + Incentive group) vs. the Control group. The secondary hypothesis is: adding incentives to the text messages is more effective for routinizing pill-taking (testing outcomes in the Incentive group vs. Message group). Outcomes from this study have the potential to greatly enhance our understanding of the barriers and facilitators of medication adherence among hypertensive patients and potentially provide evidence for a low-cost and scalable intervention to improve medication adherence in clinical practice.

This pilot RCT will also include a smaller pilot of a novel data collection method, video diaries, using the Medallia Living Lens platform. A convenience sample of 30 participants (10 from each group) will be consented and enrolled, and will be asked to upload a short video in response to structured prompts once a week for three weeks. The prompts will be geared towards experiences with the study design and interventions, and the data collected will be analyzed using the Living Lens platform.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* On anti-hypertensive medication (AH)
* Own, or have access to a phone at least five days a week throughout the duration of the intervention,
* Willing to receive study text messages

Exclusion criteria:

* Under 18 years of age
* Not approved to participate by their provider
* Not willing to use MEMS caps
* Not mentally fit to provide voluntary consent
* Already enrolled in another comparable study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Ebinger JE, Ghai I, Barajas D, Vallejo R, Blyler CA, Morales M, Garcia N, Joung S, Palimaru A, Linnemayr S. Behavioural Economics to Improve Antihypertensive Therapy Adherence (BETA): protocol for a pilot randomised controlled trial in Los Angeles. BMJ Open. 2023 Jan 25;13(1):e066101. doi: 10.1136/bmjopen-2022-066101. PMID 36697048
- [Derived] Linnemayr S, Ghai I, Palimaru A, Barajas D, Vallejo R, Blyler CA, Morales EM, De Guzman M, Joung SY, Ungar S, Ebinger JE. Impact of behavioral economics to improve antihypertensive therapy adherence, a pilot randomized controlled trial in Los Angeles. Sci Rep. 2025 Nov 4;15(1):38452. doi: 10.1038/s41598-025-94805-5. PMID 41188444
- [Derived] Ghai I, Palimaru A, Ebinger JE, Barajas D, Vallejo R, Morales M, Linnemayr S. Barriers and facilitators of habit building for long-term adherence to antihypertensive therapy among people with hypertensive disorders in Los Angeles, California: a qualitative study. BMJ Open. 2024 Jul 11;14(7):e079401. doi: 10.1136/bmjopen-2023-079401. PMID 38991671

RESULTS

PARTICIPANT FLOW:
Groups:
- Incentive Group: The Incentive group will receive the same information and text messages, but in addition have a chance of winning small, intermittent rewards for taking their medication at the time coinciding with their anchoring strategy. In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits. When the participants return for their monthly visit, the study coordinator will download their MEMS-cap data and check whether this eligibility criteria was satisfied. MEMS software can be easily customized to display this information. If the patient qualifies, s/he is invited to draw one of 3 laminated cards with numbers 0, 25, and 50 out of a bag. The client receives the corresponding amount in USD in the form of a gift card immediately after the drawing.
  Behavior Economic Incentive: In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits.
  Text Message: A key insight from BE is that people typically are initially highly motivated to change their behavior, but their enthusiasm declines over time.103 To keep the importance of routinizing pill-taking salient (i.e. high on a person's mental priority list), we will send daily text messages using a freely available web platform.
Period: Overall Study
Arm/Group | Control Group | Message Group | Incentive Group
Started | 20 | 20 | 20
Completed | 17 | 13 | 18
Not Completed | 3 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Incentive Group: The Incentive group will receive the same information and text messages, but in addition have a chance of winning small, intermittent rewards for taking their medication at the time coinciding with their anchoring strategy. In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits. When participants return for their monthly visit, the study coordinator will download their MEMS-cap data and check whether this eligibility criteria was satisfied. MEMS software can be easily customized to display this information. If the patient qualifies, s/he is invited to draw one of three laminated cards with numbers 0, 25, and 50 out of a bag. The client receives the corresponding amount in USD in the form of a gift card immediately after the drawing.
  Behavior Economic Incentive: In this group, participants will be eligible for a prize drawing if they take their medication within +/- 1 hour of the time they carry out their existing routine behavior on at least 80% of days between clinic visits.
  Text Message: A key insight from BE is that people typically are initially highly motivated to change their behavior, but their enthusiasm declines over time.103 To keep the importance of routinizing pill-taking salient (i.e. high on a person's mental priority list), we will send daily text messages using a freely available web platform.
- Total: Total of all reporting groups
Arm/Group | Control Group | Message Group | Incentive Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.34 (20.24) | 63.15 (13.46) | 60.55 (13.73) | 62.68 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 10 | 10 | 11 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 4 | 3 | 2 | 9
  White | 10 | 12 | 16 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Electronically Measured Mean Medication Adherence During Intervention
Description: The MEMS-data collected continuously over the course of the three-month intervention period will be used to calculate the primary adherence variable, which is defined as the percentage of timely (within 1 hour of anchor time) actual bottle openings out of the total number of prescribed bottle openings (# of actual once-a-day bottle openings within 1 hour of anchor time during the intervention period / # of prescribed once-a-day bottle openings during the intervention period). Only one of the anti-hypertension (AH) medications will be used to measure adherence
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Percentage of Timely Med Adherence
Arm/Group | Control Group | Message Group | Incentive Group
Number analyzed (Participants) | 20 | 20 | 20
Percentage of Timely Med Adherence | 87 (22) | 95 (34) | 92 (38)

2. Primary Outcome: Electronically Measured Mean Medication Adherence Post Intervention
Description: MEMS data will also be collected continuously over the six-month post intervention period. These data will be used to evaluate the post-intervention mean adherence, whose definition is identical to the primary outcome 1: ratio of the number of actual bottle openings to the prescribed bottle openings.
Time Frame: 6 months post intervention
Reporting Status: Not Posted, anticipated posting 2024-12

3. Primary Outcome: Routinization of AH Adherence Post-intervention
Description: This measure would be calculated as the fraction of scheduled pills taken within a one-hour window around the typical time that participants report completing their existing routine behavior that anchors their pill-taking, for all visits made post-intervention.
Time Frame: 6 months post intervention
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: Hypertension Control
Description: This is a reliable biological measure of AH adherence since controlled blood pressure is correlated with high AH medication adherence. This measure will be defined as a binary variable indicating whether or not the blood pressure measured was < 130/80 mmHg. The measure will be calculated for two time periods: at the end of the intervention and at the end of the post-intervention period.
Time Frame: 3 months and 9 months
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Control Group | Message Group | Incentive Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04029883/Prot_001.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04029883/SAP_002.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04029883/ICF_000.pdf